CLINICAL TRIAL: NCT07002892
Title: Effectiveness of Corticosteroid and 5% Dextrose Versus USG-guided Ozone Injections in Patients With Carpal Tunnel Syndrome: Three Blind Randomized Studies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunus Burak Bayır (Other Government)
Responsible Party: Sponsor-Investigator, Yunus Burak Bayır, Yunus Burak Bayır, Principal İnvestigator ,specialist doctor, Ankara Etlik City Hospital
Organization: Ankara Etlik City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024/11
Record Dates: First submitted 2025-05-25; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-11

CONDITIONS: Carpal Tunnel Syndrome Treatment
Keywords: Ozone therapy; corticosteroid injection; %5 dextrose injection; median nerve; carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Our study was designed as a prospective, triple-blind, randomized study. Patients who applied to our hospital's PMR outpatient clinic and were diagnosed with moderate carpal tunnel syndrome by EMG will be included in the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: İnvestigator, out comes assessor and participants will be blind to which procedure is performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ozon treatment group (Active Comparator): Each patient will receive 2 ml 10 μg/ml ozon perineural injection into the median nerve under US guidance, for 1 session.
  Interventions: Drug: Ozon treatment
- %5 dextrose injection group (Active Comparator): Each patient will receive 2 ml 5% dextrose perineural injection into the median nerve under US guidance, for 1 session.
  Interventions: Drug: Dextrose 5%
- corticosteroid injection group (Active Comparator): Each patient will receive 2 ml:(1 ml betamethasone dipropionate+1 ml saline) perineural injection into the median nerve under US guidance, for 1 session.
  Interventions: Drug: Steroid treatment

INTERVENTIONS:
Drug: Ozon treatment — Each patient will receive 2 ml 10 μg/ml ozon perineural injection into the median nerve under US guidance, for 1 session.
  Arms: ozon treatment group
Drug: Steroid treatment — Each patient will receive 2 ml:(1 ml betamethasone dipropionate+1ml saline) perineural injection into the median nerve under US guidance, for 1 session.
  Arms: corticosteroid injection group
Drug: Dextrose 5% — Each patient will receive 2 ml %5 dextrose perineural injection into the median nerve under US guidance, for 1 session.
  Other Names: perineural dextrose injection
  Arms: %5 dextrose injection group

SUMMARY:
Effectiveness of corticosteroid and 5% dextrose versus USG-guided ozone injections in patients with carpal tunnel syndrome: Three blind randomized studies

DETAILED DESCRIPTION:
Patients who were diagnosed with moderate CTS by EMG after clinically diagnosing CTS in our hospital's PTR clinic will be included in our study. At the beginning of the study, based on the study conducted by Wu et al. (1) who evaluated the effectiveness of dextrose prolotherapy in the treatment of patients diagnosed with carpal tunnel syndrome, the minimum number of patients required for each group was determined as 20 with a mean pain VAS change of 20%, a significance level of 0.05 and a power analysis of 95%. Considering that there may be a 20% loss during the study, it was decided to include a total of 72 patients, at least 24 patients for each group.

Patients who meet the inclusion criteria and fill out the "Informed Volunteer Consent Form" will be numbered according to their application order to the PTR clinic and will be randomized into three groups of 24 people using the "Research Randomizer" computer program, with the first group being the Ozone Group (OG), the second group being the Dextrose Group (DG) and the third group being the Corticosteroid Group (SG). Initial evaluations of the participants will be made before the injection. Each patient will receive one session of perineural injection of 1 ml betamethasone dipropionate mixed with 1 ml physiological serum to the first group; 2 ml 5% dextrose to the second group; and 2 ml 10 pg/ml ozone to the third group. The solutions to be administered will be prepared by one person in syringes that are taped shut from the outside, and then applied with a 27-gauge needle by a specialist physician who has no role in the evaluation of the results of the randomization section, from the proximal entrance of the carpal tunnel (scaphoid-psiform plane) under ultrasound guidance. In addition, each patient will wear a wrist splint for 8 hours daily during the post-treatment follow-up period. Treatment follow-up evaluations will be evaluated blindly by another specialist physician who has no role in the randomization, outcome evaluation and injection. Pre-treatment Visual Analog Scale (Global Pain), Boston Carpal Tunnel Questionnaire (Symptom Severity Scale and Functional Status Scale), Ultrasound (Measurement of median nerve cross-sectional area at pisiform level), EMG (Distal motor latency and sensory nerve conduction velocity), Hand grip strength measurement test (Dynamometer), VAS, Boston Carpal Tunnel Questionnaire, Ultrasound, Hand grip strength measurement test at the 4th week, VAS, Boston Carpal Tunnel Questionnaire, Ultrasound, Hand grip strength measurement test at the 12th week and VAS, Boston Carpal Tunnel Questionnaire, Ultrasound, Hand grip strength measurement test at the 24th week.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 years old
* Have been clinically diagnosed with carpal tunnel syndrome
* Confirmation of moderate CTS diagnosis with EMG
* Having typical CTS symptoms for at least 3 months
* Not having benefited from splinting and rest

Exclusion Criteria:

* History of polyneuropathy, brachial plexopathy, thoracic outlet syndrome or wrist surgery
* History of inflammatory arthritis, hypothyroidism, pregnancy, rheumatologic disorders or pacemaker
* Current warfarin use, previous corticosteroid injection for CTS, trauma or neoplasm at the injection site, hypersensitivity to corticosteroids or skin infection(injection site)
* G6PD deficiency, hyperthyroidism, thrombocytopenia, severe cardiovascular instability and those receiving ACE inhibitors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale(VAS) | This evaluation will be made and recorded at the baseline, at the 4th, 12th and 24th weeks after the procedure.
  Global pain:The VAS used for pain assessment consists of a line drawn in the form a ruler,and numbers from 0 to 10(with 0 as ''no pain'' and 10 as ''unbearable pain'' ) were asked to score.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Questionnaire | This evaluation will be made and recorded at the baseline, at the 4th, 12th and 24th weeks after the procedure.
  symptom severity and functional status scale
Electromyography | This evaluation will be made and recorded at the beginning and at 24th weeks
  Distal motor latency and sensory nerve conduction velocity
Dynamometer | This evaluation will be made and recorded at the baseline, at the 4th, 12th and 24th weeks after the procedure.
  Hand grip strength measurement test
Ultrasound | This evaluation will be made and recorded at the baseline, at the 4th, 12th and 24th weeks after the procedure.
  Median nerve cross-sectional area measurement at the pisiform level

CONTACTS AND LOCATIONS:
Overall Officials: BAŞAK MANSIZ KAPLAN, ASSOC. PROF., Study Chair — Ankara Etlik City Hospital; DAMLA CANKURTARAN, ASSOC. PROF., Study Chair — Ankara Etlik City Hospital; SELİN ÇELEBİER, ASSİSTANT DOCTOR, Study Chair — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forogh B, Mohamadi H, Fadavi HR, Madani SP, Aflakian N, Ghazaie F, Babaei-Ghazani A. Comparison of Ultrasound-Guided Local Ozone (O2-O3) Injection Versus Corticosteroid Injection in Patients With Mild to Moderate Carpal Tunnel Syndrome. Am J Phys Med Rehabil. 2021 Feb 1;100(2):168-172. doi: 10.1097/PHM.0000000000001546. PMID 32732745
- [Background] Elawamy A, Hassanien M, Talaat EA, Ali AM, Roushdy ASI, Kamel EZ. Intra-Carpal Injection of Ozone versus Methylprednisolone in Carpal Tunnel Syndrome of Systemic Sclerosis Patients: A Randomized Single-Blind Clinical Trial. Pain Physician. 2021 Jul;24(4):E453-E458. PMID 34213870
- [Background] Bahrami MH, Raeissadat SA, Nezamabadi M, Hojjati F, Rahimi-Dehgolan S. Interesting effectiveness of ozone injection for carpal tunnel syndrome treatment: a randomized controlled trial. Orthop Res Rev. 2019 May 6;11:61-67. doi: 10.2147/ORR.S202780. eCollection 2019. PMID 31123423
- [Background] Babaei-Ghazani A, Moradnia S, Azar M, Forogh B, Ahadi T, Chaibakhsh S, Khodabandeh M, Eftekharsadat B. Ultrasound-guided 5% dextrose prolotherapy versus corticosteroid injection in carpal tunnel syndrome: a randomized, controlled clinical trial. Pain Manag. 2022 Sep;12(6):687-697. doi: 10.2217/pmt-2022-0018. Epub 2022 Jul 18. PMID 35848821
- [Background] Nasiri A, Rezaei Motlagh F, Vafaei MA. Efficacy comparison between ultrasound-guided injections of 5% dextrose with corticosteroids in carpal tunnel syndrome patients. Neurol Res. 2023 Jun;45(6):554-563. doi: 10.1080/01616412.2022.2164453. Epub 2023 Jan 8. PMID 36617808
- [Background] Wu YT, Ke MJ, Ho TY, Li TY, Shen YP, Chen LC. Randomized double-blinded clinical trial of 5% dextrose versus triamcinolone injection for carpal tunnel syndrome patients. Ann Neurol. 2018 Oct;84(4):601-610. doi: 10.1002/ana.25332. Epub 2018 Oct 4. PMID 30187524